CLINICAL TRIAL: NCT04960566
Title: Targeting Hypervigilance and Autonomic Arousal: the Psycho-physiologic Model of GERD
Brief Title: Targeting Hypervigilance and Autonomic Arousal: the Psycho-physiologic Model of Gastroesophageal Reflux Disease (GERD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Washington University School of Medicine (Other); University of California, San Diego (Other); Vanderbilt University School of Medicine (Other)
Responsible Party: Principal Investigator, John Pandolfino, Hans Popper Professor of Medicine and Chief, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00214532; R01DK092217 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-07-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eCBT+ (Experimental): eCBT+ participants will be enrolled in 6, 45-minute sessions delivered via a secure video platform with a GI psychologist. To reinforce concepts reviewed in the sessions, participants will complete weekly home practice exercises. The targets are 1) improved maladaptive cognitive-affective processes associated with increased hypervigilance and symptom anxiety, 2) reduced behaviors associated with EHA including avoidance, increased medication/healthcare utilization and 3) reduced autonomic nervous system (ANS) arousal by increased HRV. Participants will learn to identify, question, and modify maladaptive thoughts, beliefs, and assumptions related to their symptoms (symptom anxiety). Systematic exposure to feared events are used to reduce maladaptive coping strategies (hypervigilance, PPI overuse, HCU). Specific, paced diaphragmatic breathing exercises (Resonance Frequency Breathing) designed to increase HRV are the last component (visceral hypersensitivity, reflux physiology).
  Interventions: Other: Cognitive Behavioral Therapy
- Sham-SOC Lifestyle Coaching (Sham Comparator): Patients randomized to the SOC condition will receive lifestyle guidance recommended for patients with GERD over a period of 6, 45-minute sessions with the GI psychologist to maintain consistency of delivery between the two intervention arms. Topics include maintaining a healthy weight, identifying triggering food and drink, making healthy food choices, eating behaviors, smoking and/or alcohol use, and timing of meals. The SOC condition will be carefully designed to not include any principles of the eCBT+ condition rather be based solely on patient education and encouragement to practice lifestyle changes on their own.
  Interventions: Other: Sham-SOC Lifestyle Coaching

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — The CBT intervention is based on the theoretical framework that under stress (reflux symptoms) a person makes a rapid cognitive appraisal of the potential threat (automatic thoughts), leading to both emotional and physical responses in the body, thereby reacting behaviorally (avoidance, increased HCU) in an attempt to mitigate unpleasantness. CBT is a collaborative, present-focused treatment that utilizes a skills-based approach with home practice exercises. CBT targets automatic thoughts and appraisals of threat via education, self-monitoring of stressors and symptoms, and strategies to reframe problematic thinking patterns to more adaptive ones. Resonance frequency breathing (RFB) is achieved when a person breathes at a pace, typically 4 to 6 breaths per minute, that engages the body's baroreflex to modulate arousal. Prior research demonstrates 4 to 6 weeks of RFB training is sufficient to significantly increase baseline HRV with enduring effects for up to 6 months.
  Arms: eCBT+
Other: Sham-SOC Lifestyle Coaching — Sham-SOC Lifestyle Coaching
  Arms: Sham-SOC Lifestyle Coaching

SUMMARY:
GERD affects roughly 20% of the U.S. population and the direct and indirect costs of GERD are substantial, totaling close to 50 billion dollars per year. Evidence supports that a large proportion of this cost and poor clinical outcomes in GERD are related to poor healthcare decisions by both the physician and the patient. The problem of inappropriate GERD management stems from three main issues. First, the disease is heterogeneous and requires treatment informed by a precision model. Second, the current paradigm largely ignores the important brain-gut interactions that drive symptoms and healthcare utilization. Third, there is a paucity of well-performed comparative effectiveness trials focused on assessing treatments beyond acid suppression. We will use physiomarkers defined during the previous funding cycle to phenotype the patients and use cognitive behavioral interventions to modulate hypervigilance to test the Psycho-Physiologic Model of GERD. Cognitive Behavioral Therapy (CBT) is able to improve hypervigilance and symptom specific autonomic arousal and thus, we will test our theory that CBT can improve outcomes in GERD by targeting these two important psychologic stressors. We will also continue our focus on the interplay of psychology and physiology by determining whether increased mucosal permeability is associated with reflux perception and whether this is modified by hypervigilance and autonomic disruption.

DETAILED DESCRIPTION:
OVERVIEW: In this randomized, sham-controlled phase II/III adaptive trial, we will randomize 250 subjects with symptoms of GERD to eCBT+ (esophageal Cognitive Behavioral Therapy) or sham-SOC (Standard of Care) Lifestyle Coaching. Each subject will receive 6 sessions of 45 minutes each delivered by telehealth. The study will be conducted at two institutions: Northwestern University and Washington University. The interventions will be delivered by GI Health psychologists based at Northwestern University.

RANDOMIZATION AND BLINDING: Participants will be blinded as to the intervention they will receive. Participants will be randomized in the following manner: In Aim 1, we will block on site (NU or WashU) and randomize patients to eCBT+ or SOC within sites. In Aim 2, we will block on site and whether patients have hypersensitivity. Patients within site and hypersensitivity category (no vs. yes) will be randomized. Note that in randomizing in this way, patients for Aim 3 who exhibit hypersensitivity will also be randomized within site. We will allocate participants to one of 2 study arms in a blinded fashion: eCBT+ (esophageal Cognitive Behavioral Therapy) or sham-SOC Lifestyle Coaching. Subjects will be de-briefed at their week 25 visit.

STUDY PROCEDURES: Study procedures include mucosal impedance (MI) performed during standard of care endoscopy, the use of questionnaires: GERD PROMIS (a measure of symptoms), EHAS (Esophageal Hypervigilance and Anxiety Scale), NEQOL (Northwestern Esophageal Quality of Life), GERDQ (a measure of symptom frequency), and patient satisfaction, as well as measurement of heart rate variability both at the research site and via continuous FitBit usage throughout the treatment period. For Aim 3, repeat endoscopy, mucosal impedance, and pH impedance will be performed on a subset of patients 8 weeks after conclusion of intervention.

ENDPOINTS: Primary endpoints include change in symptoms and quality of life as measured by GERDQ, GERD PROMIS and NEQOL questionnaires, change in hypervigilance and symptom-specific anxiety as measured by EHAS and change in autonomic arousal as measured by HRV before and after treatment with either intervention arm. Secondary endpoints include change in mucosal impedance measurements and symptom index (as determined by pH-Impedance monitoring) before and after treatment, as well as patient satisfaction with treatment and engagement with treatment as defined by the number of sessions completed.

RATIONALE: We selected a parallel design study to explore the treatment effect of eCBT+ compared to a sham-SOC Lifestyle Coaching approach. Power and sample size considerations were based on the primary aim of comparing questionnaire results and HRV measurements in the proposed two-arm clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects (females of childbearing potential should be on highly effective contraceptive methods)
* Aged 18-80 years old
* Mentally capable to provide informed consent
* Fluent in English
* Have symptoms of GERD (heartburn, regurgitation, and non-cardiac chest pain)
* Have failed an appropriate compliant trial of PPI therapy with a GERDQ score ≥6.
* Able to undergo endoscopy, ambulatory reflux monitoring, and manometry
* Be interested in behavioral interventions for ongoing symptoms.

Exclusion Criteria:

* Participation in a concurrent clinical trial or completed another trial within past 8 weeks.
* Active severe erosive esophagitis (Los Angeles Grade C or D), Long segment Barrett's esophagus (Zap score of 4)
* Prior gastrointestinal surgery of the esophagus and/or stomach
* Current signs or symptoms of heart disease. All patients with non-cardiac chest pain are required to have a cardiologist evaluation as standard of care work up in the evaluation of non-cardiac chest pain.
* Unstable medical illness with ongoing diagnostic work-up and treatment. Patients with well-controlled hypertension, diabetes and a remote history of ischemic heart disease that is deemed stable, as judged by the investigator can be included.
* History of drug addiction, drug abuse or alcoholism.
* Current neurologic or cognitive impairment, which would preclude ability to obtain informed consent.
* Pregnant patients.
* Special vulnerable populations including children, prisoners, institutionalized individuals.
* Bleeding disorder or requirement of NSAID/aspirin during monitoring period.
* Drugs that affect gastrointestinal symptoms (H2 blockers, antacids, metoclopramide, domperidone, erythromycin, anticholinergics [bentyl, levsin, belladonna etc.]). Antidepressants can be continued at stable dose.
* Patients found to have achalasia, a spastic disorder, hypercontractile disorder or functional obstruction at the esophagogastric junction will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
GERD PROMIS | Week 9
  25-item measure of GERD symptom severity rated on Likert scale across 4 domains. Higher scores denote more GERD symptoms.
GERD PROMIS | Week 25
  25-item measure of GERD symptom severity rated on Likert scale across 4 domains. Higher scores denote more GERD symptoms.
NEQOL | Week 9
  14-item measure of HRQoL related to esophageal symptoms, rated on Likert scale. Higher scores denote greater negative impacts on HRQoL.
NEQOL | Week 25
  14-item measure of HRQoL related to esophageal symptoms, rated on Likert scale. Higher scores denote greater negative impacts on HRQoL.
EHAS | Week 9
  15-item measure of esophageal hypervigilance and symptom specific anxiety rated on Likert scale. Higher scores indicate more hypervigilance and anxiety.
EHAS | Week 25
  15-item measure of esophageal hypervigilance and symptom specific anxiety rated on Likert scale. Higher scores indicate more hypervigilance and anxiety.
Variation in Heart Rate Variability (HRV) | from the date of randomization through the treatment period, up to 9 weeks
  HRV will be measured using the time domains RMSSD and pNN50 calculated at each time point, as well as daily averages throughout treatment period.
Heart Rate Variability (HRV) | Week 9
  HRV will be measured using the time domains RMSSD and pNN50 calculated at each time point, as well as daily averages throughout treatment period.
Heart Rate Variability (HRV) | Week 25
  HRV will be measured using the time domains RMSSD and pNN50 calculated at each time point, as well as daily averages throughout treatment period.
Esophageal Permeability | Week 9
  Permeability will be measured utilizing Mucosal Impedance (MI) measurement. Higher MI value indicates lower permeability
Symptom Index | Week 9
  Symptom index is defined as the number of symptoms associated with reflux divided by the total number of symptoms as determined by pH-Impedance

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire - 8 | Week 9
  8-item measure of patient satisfaction with treatment rated on Likert scale. Higher scores indicate greater satisfaction with treatment.
Sessions completed | Week 9
  Number of sessions of intervention (either arm) completed by each subject. Higher number of sessions indicate greater engagement with treatment

CONTACTS AND LOCATIONS:
Overall Officials: John E Pandolfino, MD, Principal Investigator — Northwestern University; Tifffany Taft, PsyD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No